CLINICAL TRIAL: NCT06328543
Title: Repetitive Applications of Pruritogens and Effects of a Cutaneous-induced Pain Stimulation on Nonhistaminergic Itch Perception
Brief Title: Itch Sensation Induced by Multiple Applications of Pruritogens (temporal Summation)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20210046 4th project
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Histamine; Cowhage
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Intervention Model Description: The participants will randomly receive applications of cowhage and histamine
Who Masked: Participant
Masking Description: Participant will be blinded about application of pruritogens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1st pruritogen (Experimental): The subproject is conducted in 1 session (approx. 3 hours in total) divided into two parts. In the first part, 3 test areas (3x3 cm) will be selected on one forearm of the subject. The 3 areas will be randomly treated with 1 application of cowhage, 2 applications of cowhage (the second application will be conducted 90 seconds after the first one in the same area), and 2 applications of cowhage (the second application will be conducted 180 seconds after the first one in the same area). Itch will be monitored using a VAS (visual analog scale) for 15 min in each session. After the removal of cowhage, FLPI, alloknesis, and mechanically evoked itch will be measured.
  Interventions: Other: Histamine
- 2nd pruritogen (Experimental): The second part will be conducted 20 minutes after the first part, and the procedure will be the same, but using histamine instead of cowhage. The two parts will be randomized between subjects.
  Interventions: Other: Cowhage

INTERVENTIONS:
Other: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine.
  Arms: 1st pruritogen
Other: Cowhage — 25 spicules will be inserted in the center of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration.
  Arms: 2nd pruritogen

SUMMARY:
In This experiment, the investigators would like to design a new itch model based on the temporal summation of pruritic stimuli. The hypothesis behind this study (temporal summation) is that two overlapped applications of pruritogens will result in a higher itch sensation compared with a single application.

DETAILED DESCRIPTION:
Chronic itch affects approximately a fifth of the global population and is associated with substantial negative consequences for the affected individuals. Furthermore, there is a lack of efficient treatment options for chronic itch. In order to mimic a clinical itch condition as presented in patients, the aim of the project is to investigate a new itch model based on the multiple applications of pruritogens (temporal summation). In particular, the purpose is to evaluate if a single application of cowhage/histamine (non-histaminergic and histaminergic itch, respectively) results in a lower itch sensation compared with two overlapped applications of the pruritogens on the same area.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand Englis

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis), musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder, or mental illnesses that may affect the results
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids
* Skin diseases (e.g. atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of itch | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'

SECONDARY OUTCOMES:
Microvascular reactivity | 10 minutes after every itch inductions
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Alloknesis | 12 minutes after every itch inductions
  Alloknesis sensation is measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.
Mechanically evoked itch | 15 minutes after every itch inductions
  Mechanically evoked itch is measured using three von Frey filaments of 4.08, 4.16 and 4.31 (1.0, 1.4, 2.0 g, respectively) (North Coast Medical, Gilroy, CA). The center of the skin area is stimulated by 3 pricks, repeated 3 times in short succession. After a total of 9 stimulations, the participants will report the itch elicited on a numerical rating scale (NRS) from 0 to 10 (0 = "no itch"; 10 = "worst imaginable itch").

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No